CLINICAL TRIAL: NCT05615376
Title: Beat to Beat A Prospective Study in Paediatric, Adolescent and Young Adult Patients Aged 7 to 18 Years of Age Who Are Undergoing or Have Undergone Cancer Therapy to Evaluate the Agreement Between QTc Measured Using 12 Lead Electrocardiogram (ECG) and a Wearable Device ECG
Brief Title: Beat to Beat A Study in Paediatric, Adolescent and Young Adult Patients Who Are Undergoing or Have Undergone Cancer Therapy to Evaluate the Agreement Between QTc Measured Using 12 Lead Electrocardiogram (ECG) and a Wearable Device ECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 88476
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms; Cardiac Arrhythmia
Keywords: QT prolongation; cancer; paediatric; ECG application; 12 lead ECG
MeSH Terms: conditions — Neoplasms; Arrhythmias, Cardiac; Long QT Syndrome | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ECG App arm (Experimental): Participants will be provided with a wearable device on Day 1 and Day 4 whilst admitted in hospital.
  Interventions: Device: ECG application; Device: 12 lead ECG

INTERVENTIONS:
Device: ECG application — The app together with the wearable device will record a V1 (Left wrist) or V2 (left ankle) ECG reading. These measurements will be conducted on Day 1 and Day 4.
Device: 12 lead ECG — The 12 lead ECG will measure corrected QT interval by recording RR and QT intervals on Day 1 and Day 4. This will be performed within the same episode of care as the wearable device ECG recording. There is no need to perform both at exactly the same time point, but within a 15 minute window.

SUMMARY:
A prospective study in paediatric, adolescent and young adult patients aged 7 to 18 years to evaluate the agreement between QTc measured using 12 lead electrocardiogram (ECG) and the wearable device ECG.

DETAILED DESCRIPTION:
Rationale: Leveraging existing wearable technology has the ability to scale routine screening strategies across large populations and can facilitate ambulatory care. In recent years, wearable technology has rapidly diffused into consumer markets and provides unique opportunities to engage individuals on health issues of personal interest, and to collect personal health data. One example of such technology is the ability to perform electrocardiogram (ECG) type traces on wearable devices. However, utilization of this data source to improve patient outcomes has not been fully realized in the health care field. An app-based heart ECG algorithm that can be remotely analysed for QTc prolongation with potential to then notify the user of such potential irregularities could lead to widespread screening, detection and initiation of treatment solutions (i.e. correction of electrolytes, alteration of exacerbating medications, cardiac monitoring etc).

Trial Design: This will be a prospective, single arm, experimental, non-significant risk study conducted with the assistance of eligible participants. Parents or mature minors will download the Beat to Beat app, once consented.

Once consented the wearable device will be paired to the parent/guardians phone following the steps provided by the wearable device app. Once the device is paired and the study coordinator has assisted with the download of 'Beat to Beat' app, the patients will then be able to commence the ECG readings. A 12 lead ECG will be performed by the study team and immediately following this, an ECG will be recorded on the wearable device. The wearable device will be placed on the left wrist for a Lead I reading, on the left lower abdomen for a Lead II reading and in the fourth intercostal space left parasternal for a chest V2 Lead reading. Recording of the 12 lead ECG and wearable device ECG will be repeated again 4 days later. Once both timepoints (and two device recordings for each time period) have been completed the ECGs will be retrieved from the Beat to Beat app. Both the 12 lead and wearable device ECG will be de-identified and given a patient identifier before being uploaded into the REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric or adolescent diagnosis of cancer AND an inpatient of The Royal Children's Hospital, Melbourne for at least 5 days at the time of consent.
* Patient age ≥ 7 years at time of eligibility screening
* If age < 18 years, parent or guardian able to provide consent
* Parental or participant ( if > 18 years of age) possession of the following at time of eligibility screening, ascertained from automatic hardware/software/device pairing check:

  1. iPhone (6s or later) with iOS version 15.0 or later defined as iPhone model/iOS version used to complete screening eligibility.
  2. Proficient in written and spoken English, defined by self-report of comfort reading, writing, and speaking English on iPhone.
  3. Valid phone number associated with iPhone, ascertained from self-report.
  4. Valid email address, ascertained from self-report.
  5. Participants or parents need to be able to press down on the wearable device crown for 30 seconds

Exclusion Criteria:

* Unable to wear the wearable device.
* < 18 years of age without guardian or parent to provide consent.
* Interpreter required for consent purposes.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Recording of a 12 lead ECG and wearable device ECG | Day 1 of inpatient stay
  12 lead ECG and wearable device ECG recordings will be taken at the time point of care. The wearable device ECG will be placed on the left wrist to record a V1 (lead I) ECG and on the left ankle to record a V2 (lead II) ECG reading from which the QT interval can be calculated.
Recording of a 12 lead ECG and wearable device ECG | Day 4 of inpatient stay
  12 lead ECG and wearable device ECG recordings will be taken at the time point of care. The wearable device ECG will be placed on the left wrist to record a V1 (lead I) ECG and on the left ankle to record a V2 (lead II) ECG reading from which the QT interval can be calculated.
Calculation of QT interval by two blinded health professionals | Day 1 of inpatient stay
  The wearable device ECG and 12 lead ECG will be de-identified and given appropriate study numbers. This data will be listed separately for each patient. The QT interval for each recording will be calculated. This is the time corresponding to beginning of depolarization to repolarization of the ventricles. It is calculated using a standardised approach (Fridericia's formula:QTcF = QT divided by cube root of RR).
Calculation of QT interval by two blinded health professionals | Day 4 of inpatient stay
  The wearable device ECG and 12 lead ECG will be de-identified and given appropriate study numbers. This data will be listed separately for each patient. The QT interval for each recording will be calculated. This is the time corresponding to beginning of depolarization to repolarization of the ventricles. It is calculated using a standardised approach (Fridericia's formula:QTcF = QT divided by cube root of RR).

SECONDARY OUTCOMES:
Number of Participants with Abnormal QTc that is greater than 0.48mm on 12 lead ECG and wearable device ECG | Day 1 inpatient stay
  From the analysis of QT measurements from Outcome 2, prolonged or abnormal QTc measurement will be noted. An abnormal QTc is greater than 0.48mm. This data will be collected separately for each patient.
Number of Participants with Abnormal QTc that is greater than 0.48mm on 12 lead ECG and wearable device ECG | Day 4 inpatient stay
  From the analysis of QT measurements from Outcome 2, prolonged or abnormal QTc measurement will be noted. An abnormal QTc is greater than 0.48mm. This data will be collected separately for each patient.
Sensitivity calculations of wearable device vs 12 Lead ECG | Day 1 inpatient stay
  Sensitivity is calculated only in the participants who are declared to have QTc prolongation (abnormal QTc) and is calculated as the proportion patients with QTc prolongation on the wearable device among those with QTc prolongation on the 12-lead ECG.
Sensitivity calculations of wearable device vs 12 Lead ECG | Day 4 inpatient stay
  Sensitivity is calculated only in the participants who are declared to have QTc prolongation (abnormal QTc) and is calculated as the proportion patients with QTc prolongation on the wearable device among those with QTc prolongation on the 12-lead ECG.
Specificity calculations of wearable device vs 12 Lead ECG | Day 1 inpatient stay
  Specificity is calculated only in participants who do not have QTc prolongation and is calculated as the proportion patients who do not have QTc prolongation on the wearable device among those who do not have QTc prolongation on the 12-lead ECG.
Specificity calculations of wearable device vs 12 Lead ECG | Day 4 inpatient stay
  Specificity is calculated only in participants who do not have QTc prolongation and is calculated as the proportion patients who do not have QTc prolongation on the wearable device among those who do not have QTc prolongation on the 12-lead ECG.
To calculate the interobserver variability between the two health care professional readings of QTc. | Day 1 inpatient stay
  The corrected QT interval will be calculated on both the wearable device ECG and the 12 lead ECG for each patient and measured by a health professional. QT interval will be calculated by the health professional by using the QT and RR interval from the ECGs using Frederichia's interval (QTcF = QT divided by cube root of RR). This data will be collected separately for each patient. The standard deviation of the difference in QTc interval between the two observers will be reported.
To calculate the interobserver variability between the two health care professional readings of QTc. | Day 4 inpatient stay
  The corrected QT interval will be calculated on both the wearable device ECG and the 12 lead ECG for each patient and measured by a health professional. QT interval will be calculated by the health professional by using the QT and RR interval from the ECGs using Frederichia's interval (QTcF = QT divided by cube root of RR). This data will be collected separately for each patient for each patient The standard deviation of the difference in QTc interval between the two observers will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Rachel Conyers, Principal Investigator — The Royal Children's Hospital/Murdoch Children's Research Institute
Locations (1):
- The Royal Children's Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the Beat to Beat trial will be available 12 months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified data set collected for the analysis of the trial will be available for six months after publication of the primary outcome. The study protocol can be obtained from Murdoch Children's Research Institute. Prior to access to any data the following would be required: a data access agreement must be signed by all relevant parties, the investigators of the study must see and approve the analysis plan describing how the data will be analysed. There must be also an agreement around appropriate acknowledgement in any future publications.
Access Criteria: The data may be obtained from the Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au
URL: https://www.melbournechildrens.com/mctc/